CLINICAL TRIAL: NCT02966314
Title: A Phase IV, Randomized, Double-Blind, Placebo-Controlled Exploratory Study of Xolair (Omalizumab) for Treatment of Idiopathic Angioedema in Patients Who Remain Symptomatic Despite Current Therapy
Brief Title: Treatment of Idiopathic Angioedema With Xolair as Add-on Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-0645; SMPH/MEDICINE/MEDICINE*A (Other: UW Madison); A534220 (Other: UW Madison); Protocol Version 5/22/2018 (Other: UW Madison)
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Results first posted 2021-11-22 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Idiopathic Angioedema
Keywords: Angioedema; Idiopathic Angioedema; IAE
MeSH Terms: conditions — Angioedema | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo contains sodium chloride 0.9% and will be provided by Novartis. Placebo will be administered as a subcutaneous injection.
  Interventions: Drug: Placebos
- Omalizumab (Active Comparator): Omalizumab is a sterile, white, preservative-free, lyophilized powder, contained in a single-use vial that will be reconstituted with sterile water for injection (SWFI), USP, and administered as a subcutaneous injection. Each omalizumab vial contains 202.5 mg of omalizumab, 145.5 mg sucrose, 2.8 mg L-histidine hydrochloride monohydrate, 1.8 mg L-histidine, and 0.5 mg polysorbate 20. Each vial is designed to deliver 150 mg of omalizumab in 1.2 mL after reconstitution with 1.4 mL SWFI, USP.
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — Omalizumab 300mg subcutaneous injection once monthly for 6 months. Total dose will be divided into two 150mg/1.2mL injections.
  Other Names: Xolair
  Arms: Omalizumab
Drug: Placebos — Placebo Group (Sodium Chloride 0.9%) two 1.2mL subcutaneous injections once monthly for 6 months.
  Arms: Placebo

SUMMARY:
The overall hospitalizations for a diagnosis of angioedema doubled from the year 2000 to 2009. Although some of the cases represented hereditary angioedema or ace-inhibitor induced angioedema, the majority of episodes were idiopathic. Idiopathic Angioedema (IAE) can be life- threatening especially when affecting tissues within the respiratory tract. No clear guidelines exist for management of this important condition for clinicians. Current therapies typically include avoidance of potential triggers and use of medications either for prophylaxis or for acute events, such as antihistamines, corticosteroids, and epinephrine. There remains a critical need for therapeutic options to provide more effective prophylaxis.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, parallel group trial which will study the effects of omalizumab on patients with 2 or more episodes of Idiopathic Angioedema (IAE) in the past 6 months, despite current therapy. This study has three periods; screening, treatment, and follow-up. Subjects in the screening period will be consented and screened for eligibility criteria. 40 qualified individuals will enter the treatment period. Individuals will be randomized to either monthly subcutaneous administration of omalizumab 300mg (20 subjects) versus monthly placebo injection (20 subjects) in addition to their previously prescribed management plan for a total of 6 months. Individuals will then enter a follow-up period of 4 months. Study visits will occur monthly during the treatment period for update of clinical status and administration of omalizumab/placebo injection. After, the treatment period individuals will be seen twice for follow-up period. The entire study will consist of 10 study visits and will last approx. 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults or adolescents who are 18 years or older at the time of screening with physician diagnosis of idiopathic angioedema
* Minimum of two episodes of idiopathic angioedema in the past 6 months at the time of screening
* Management of idiopathic angioedema with a stable controller treatment plan for the prior 6 months
* Complement profile (C1 Esterase inhibitor panel) within normal reference values
* If a woman is of child-bearing potential, she must agree to a reliable form of birth control including: abstinence, oral contraceptives (birth control pills), Depo-provera, an intrauterine device (IUD), or double-barrier contraception (partner using condom and participant using diaphragm, contraceptive sponge or cervical cap, and spermicidal)

Exclusion Criteria:

* Diagnosis of Hereditary Angioedema (HAE), Acquired Angioedema, or Ace-inhibitor associated angioedema, which are forms of angioedema with known mechanisms and alternate treatment options
* Chronic Urticaria (itching and/or hives) with or without Angioedema which are known mast cell mediated processes previously shown to be responsive to the use of omalizumab
* Previous usage of omalizumab in the last 3 months which can affect the patient-related outcomes and biomarker assessments if not "washed out" of the system
* Patients, who in the judgment of the investigator, have a history or condition that might compromise patient safety or compliance, interfere with evaluations, or preclude completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Mathur, MD/PhD, Principal Investigator — UW Madison; Ravi Viswanathan, MD, Principal Investigator — UW Madison
Locations (1):
- UW Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goswamy VP, Lee KE, McKernan EM, Fichtinger PS, Mathur SK, Viswanathan RK. Omalizumab for treatment of idiopathic angioedema. Ann Allergy Asthma Immunol. 2022 Nov;129(5):605-611.e1. doi: 10.1016/j.anai.2022.07.017. Epub 2022 Jul 30. PMID 35914662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened and enrolled at the University of Wisconsin-Madison Allergy and Asthma Clinical Research Unit from March 2017 to April 2019.
Pre-assignment Details: Two participants were screened and enrolled but not randomized to an arm to start the study.
Period: Overall Study
Arm/Group | Placebo | Omalizumab
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Two participants enrolled onto the study were screened but not randomized to an arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Omalizumab | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 53 [24 to 72] | 53.8 [42 to 68] | 53.4 [24 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Height [Mean (Full Range); unit: centimeters] | 171.18 [154.9 to 185] | 180.86 [169.3 to 195.4] | 176.02 [154.9 to 195.4]
Weight [Mean (Full Range); unit: kg] | 93.4 [48.6 to 134.7] | 91.2 [54.1 to 132.2] | 92.3 [48.6 to 134.7]
Number of IAE Episodes in past 6 months [Mean (Full Range); unit: IAE Episodes] — Idiopathic Angioedema (IAE)
  IAE Episodes | 15.2 [2 to 35] | 10.6 [8 to 12] | 12.9 [2 to 35]
Duration of IAE Episodes [Mean (Full Range); unit: hours] — Average number of hours that each IAE event lasted over the previous month, as reported by participant at baseline
  hours | 14.3 [2 to 36] | 21.1 [6 to 48] | 17.7 [2 to 48]
Number of Urgent Care / Emergency Department Visits in past 6 months [Mean (Full Range); unit: visits] | 0.6 [0 to 3] | 0.2 [0 to 1] | 0.4 [0 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Mean 7-day Angioedema Activity Score (AAS7)
Description: The AAS7 Score is a measure of the frequency and intensity of angioedema episodes. The total possible range of scores over 7 days is 0-15 (mean day sum score) where higher scores indicate increased angioedema activity.
Time Frame: baseline to end of treatment period at 6 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 5 | 5
score on a scale
  baseline (2 weeks prior to randomization) | 2.8 [0 to 9] | 1.6 [0 to 4]
  6 months | 0.69 [0 to 1.75] | 0.20 [0 to 1]

2. Primary Outcome: Presence of a 7-day Angioedema Activity Score (AAS7) Greater Than 0 Across All Treatment Visits
Description: as for outcome 1
Time Frame: across all visits during treatment period (up to 6 months)
Measure: Count of Units; unit: participant visits
Units Other Than Participants: participant visits
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 5 | 5
Number analyzed (participant visits) | 103 | 120
participant visits | 38 | 4
Statistical Analysis 1: Comparison: Placebo vs Omalizumab; Test type: Superiority; p = 0.003, Regression, Logistic; Accounting for repeated measures; Odds Ratio (OR) = 18.7, 95% CI 2-sided [2.77 to 126.47]

3. Secondary Outcome: Mean Angioedema Quality of Life (AE-QoL) Questionnaire
Description: The AE-QoL Questionnaire is a 17-item survey, the total possible range of scores is transformed to a scale of 1-100 where higher score indicate increased impairment.
Time Frame: baseline to end of treatment period at 6 months
Population: 1 participant in the placebo arm was lost to follow up at the 6 month measure, but was able to be analyzed for the Primary Outcome
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 5 | 5
score on a scale
  baseline (2 weeks prior to randomization) | 28.25 [4.41 to 42.65] | 21.47 [0 to 42.65]
  6 months: number analyzed (Participants) | 4 | 5
  6 months | 19.12 [2.94 to 35.29] | 8.53 [0 to 23.53]

4. Secondary Outcome: Mean Angioedema Quality of Life (AE-QoL) Questionnaire Across All Treatment Visits
Description: as for outcome 3
Time Frame: across all visits during treatment period (up to 6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: participant visits
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 5 | 5
Number analyzed (participant visits) | 28 | 30
score on a scale | 19.0 (12.9) | 8.5 (10.4)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab; Test type: Superiority; p = 0.03, Regression, Linear; Mean Difference (Final Values) = 9.43, 95% CI 2-sided [1.24 to 17.63]

5. Secondary Outcome: Mean Visual Analog Scale
Description: The effect of treatment compared to placebo on the change in IAE severity from baseline to the end of the treatment period as recorded on a 0-100 visual analog scale. Lower numbers indicate increased severity.
Time Frame: baseline to end of treatment period at 6 months
Population: as for outcome 3
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 5 | 5
score on a scale
  baseline (2 weeks prior to randomization) | 91 [70 to 100] | 84 [30 to 100]
  6 months: number analyzed (Participants) | 4 | 5
  6 months | 88.75 [65 to 100] | 97 [85 to 100]

6. Secondary Outcome: Presence of Visual Analog Scale Less Than 100 Across All Treatment Visits
Description: as for outcome 5
Time Frame: across all visits during treatment period (up to 6 months)
Measure: Count of Units; unit: participant visits
Units Other Than Participants: participant visits
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 5 | 5
Number analyzed (participant visits) | 28 | 30
participant visits | 17 | 4
Statistical Analysis 1: Comparison: Placebo vs Omalizumab; Test type: Superiority; p = 0.03, Regression, Logistic; Accounting for repeated measures; Odds Ratio (OR) = 32.8, 95% CI 2-sided [1.49 to 720.54]

7. Secondary Outcome: Mean Number of IAE Episodes 2 Weeks Prior to Randomization
Description: Idiopathic angioedema (IAE) refers to episodes of angioedema without urticaria for which no explanation can be found despite a thorough investigation. Patients are sometimes referred to as having IAE while further investigations are being performed, and therefore this term does not necessarily represent a distinct condition, but rather a diagnostic challenge in which the pathway of swelling is yet to be determined.
Time Frame: baseline to end of treatment period at 6 months
Population: as for outcome 3
Measure: Mean (Full Range); unit: episodes
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 5 | 5
episodes
  baseline (2 weeks prior to randomization) | 1 [0 to 4] | 0.4 [0 to 1]
  6 months: number analyzed (Participants) | 4 | 5
  6 months | 0.5 [0 to 1] | 0.2 [0 to 1]

8. Secondary Outcome: Number of IAE Events Across All Treatment Visits
Time Frame: across all visits during treatment period (up to 6 months)
Measure: Mean (Standard Deviation); unit: count of events
Units Other Than Participants: participant visits
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 5 | 5
Number analyzed (participant visits) | 28 | 30
count of events | 1.8 (2.3) | 0.2 (0.5)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab; Test type: Superiority; p = 0.005, Regression, Linear; Accounting for multiple measures, using poisson distribution with natural log link; Risk Ratio (RR) = 6.9, 95% CI 2-sided [1.9 to 25.3]

9. Secondary Outcome: Change in Duration of IAE Episodes
Description: Duration of IAE Episodes is participant reported for the 6 months prior to study (baseline) and again at the 6 month time point for the time on study.
Time Frame: baseline to end of treatment period at 6 months
Population: as for outcome 3
Measure: Mean (Full Range); unit: hours
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 5 | 5
hours
  baseline (2 weeks prior to randomization) | 14.3 [2 to 36] | 21.1 [6 to 48]
  6 months: number analyzed (Participants) | 4 | 5
  6 months | 3.25 [0 to 7] | 0.5 [0 to 2.5]

10. Secondary Outcome: Number of Participants Who Visited Urgent Care or Emergency Room
Description: Count of participants who visited urgent care or the emergency room is participant reported. The baseline measure is for the 6 months prior to study, at the 6 month time point for the time on study, and the 9 month time point for the previous 3 months on study.
Time Frame: baseline, end of treatment period at 6 months, follow up at 9 months
Population: Data not collected due to study communications.
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants Who Used Rescue Medication or Corticosteroids
Time Frame: baseline, end of treatment period at 6 months, follow up at 9 months
Population: Data not collected due to study communications.
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Times Rescue Medications Were Used During the Treatment Period
Time Frame: up to 26 weeks
Measure: Count of Units; unit: instances of rescue medication use
Units Other Than Participants: instances of rescue medication use
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 5 | 5
Number analyzed (instances of rescue medication use) | 32 | 8
instances of rescue medication use
  Number of times Rescue Systemic Steroid used | 5 | 0
  Number of times rescue H1-antagonist used | 13 | 7
  Number of times rescue H2-antagonist used | 14 | 1

ADVERSE EVENTS:
Time Frame: up to 9 months
Arm/Group | Placebo | Omalizumab
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5) | Omalizumab (N=5)
Delayed Injection Site Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT02966314/Prot_SAP_000.pdf